CLINICAL TRIAL: NCT07183397
Title: Impact of Fluid Resuscitation on Venous Congestion in Cardiac Critically-ill Patients
Acronym: VExUS-CS
Status: Not yet recruiting | Type: Observational
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Pedro D. Wendel Garcia, Dr.med., Medical University of Vienna
Other Study IDs: 1706/2025
Record Dates: First submitted 2025-09-14; First posted 2025-09-19 (Actual); Last update posted 2025-09-19 (Actual); Status verified 2025-09

CONDITIONS: Cardiac and Aortic Surgery; Cardiac Anaesthesia; Venous Congestion; Fluid Resuscitation
MeSH Terms: conditions — Hyperemia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood Samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: VExUS & Cardiac Ultrasound — The VExUS system provides a semi-quantitative assessment of systemic venous congestion by integrating ultrasound evaluations of the inferior vena cava diameter, hepatic vein flow, portal pulsatility, and renal venous flow, offering a practical and comprehensive bedside tool

SUMMARY:
The objective of this study is to assess how fluid resuscitation, in the context of fluid responsiveness, affects the incidence and progression of systemic venous congestion in critically ill cardiac patients. Additionally, the study aims to evaluate the impact on clinical outcomes, with a particular focus on acute kidney dysfunction. This assessment will utilize the VExUS score in conjunction with comprehensive bedside echocardiographic evaluations.

ELIGIBILITY:
Inclusion Criteria:

* Age above 18 years
* Admission to cardiac intensive care unit

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Cardiac critically ill patients (mainly post cardiac surgery)
Sampling Method: Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2025-09-15 (Estimated); Primary Completion 2027-09 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Venous congestion | 7 days
  Venous congestion as assessed by the VExUS score at ICU admission, and on each of the first seven postoperative days.
Acute kidney injury | Twenty-eight days
  Acute kidney injury (AKI), defined through the KDIGO criteria, within seven and twenty-eight days of ICU admission.

IPD SHARING:
Plan to Share IPD: Undecided
Data is available upon reasonable request and after the approval of the Steering Committee members.